CLINICAL TRIAL: NCT05817448
Title: The Possible Role of Hypoxia-induced Autophagy and Matrix Metalloproteinase-9 in the Pathogenesis of Morbidly Adherent Placenta.
Brief Title: Hypoxia-induced Autophagy in the Pathogenesis of MAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermeen Bahaa El Dien Mohamed Ahmed, Demonstrator at Physiology department, Assiut University
Other Study IDs: hypoxia in MAP
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hypoxia; Autophagy; Placenta; Morbidly Adherent Placenta
Keywords: HIF1α; hypoxia-induced autophagy; LC3B; invasion-related markers; MMP-9; Morbidly Adherent Placenta
MeSH Terms: conditions — Hypoxia; Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: 40 pregnant women with normal placentation having no pregnancy related disorders according to the physical examination and laboratory findings.
  Interventions: Diagnostic Test: HIF 1α and LC3B expression and MMP-9 level
- placenta previa group: 40 pregnant women that will be diagnosed according to the ultrasound diagnostic criteria.
  Then according to the histopathological examination, placenta previa group will be subdivided into 2 groups, placenta previa with MAP and placenta previa without MAP
  Interventions: Diagnostic Test: HIF 1α and LC3B expression and MMP-9 level

INTERVENTIONS:
Diagnostic Test: HIF 1α and LC3B expression and MMP-9 level — 5ml of venous blood samples will be taken from all participants at 28-40 weeks of gestation for detcetion of MMP-9 level by Enzyme-Linked Immune Sorbent Assay (ELISA) kit.
  Placental tissue sample in the maternal surface will be taken during CS in placenta previa group and similar location in maternal surface will be sampled after placental delivery in control group for histopathology and immunohistochemistry for detection of HIF 1α and LC3B expression

SUMMARY:
To investigate the role of HIF 1α and LC3B in the pathogenesis of MAP, to evaluate the role of MMP-9 in the antenatal prediction of MAP, and to compare the expression of HIF1α, LC3B, and level MMP-9 between patients of placenta previa with MAP and patients with normal placentation.

DETAILED DESCRIPTION:
Cesarean section (CS) rate has been rising rapidly in the recent years.One of the complications of repeated CS is placenta previa, an implantation of placenta on or near internal os.

Morbidly adherent placenta (MAP), known also as placenta accreta spectrum, has histopathologic and clinical types. The placenta becomes abnormally adherent to the uterine wall, fails to separate leading to massive blood loss and possible hysterectomy. The risk of MAP in patient with placenta previa increases with repeated CS.

Theories for development of MAP include abnormal trophoblastic invasion of myometrium, abnormal decidualization, neovascularization and reduction of apoptosis of trophobalsts.

In early pregnancy: the trophoblasts invade spiral arteries and reduce blood flow to the placenta 00leading to hypoxia. Hypoxia inducible factor 1 alpha (HIF-1α), a protein involved in cellular adaptation to hypoxia, increases throughout pregnancy and contributes in the invasion of trophoblasts. Excessive invasion in MAP might prolong the hypoxia, increasing the expression of HIF1α.

Autophagy is a process for managing and removing the damaged organelles and cellular proteins in hypoxia. It supports the trophoblasts. Hypoxia induced autophagy markers such as LC3B might be enhanced by MAP.

Matrix metalloproteinase-9 (MMP-9) plays an important role in cell invasion and placental implantation. Disturbance of MMP-9 might alter the trophobalsts invasion resulting in MAP .

The investigators hypothesize that hypoxia, autophagy and invasiveness are linked to the pathophysiology of MAP, so we will assess the expression of HIF1α, LC3B to estimate their role beside MMP-9.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age: more than 28 weeks up to 40 weeks.
2. Pregnant women with at least one previous CS.
3. Singleton pregnancy.
4. Patient known to have placenta previa by 2D ultrasound.
5. Heamodynamically stable patient.

Exclusion Criteria:

1. Multiple pregnancy.
2. Gestational age less than 28 weeks.
3. Heamodynamically unstable patient.
4. Hypertensive disorder with pregnancy.
5. Gestational diabetes.
6. IUGR.
7. Patient with bleeding tendency or using anticoagulant.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: selected from out patient's clinic of the department of Obstetrics and Gynecology at Assiut University Hospital, Assiut, Egypt,
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Compare the expression of HIF 1α and LC3B by immunohistochemistry and the level of MMP-9 | 28-40 weeks of gestation.
  To explore the mechanism of abnormal trophoblasts invasion in MAP.

SECONDARY OUTCOMES:
Measure MMP-9 concentration in the maternal plasma | 28-40 weeks of gestation.
  To verify its usefulness as an antenatal predictor of MAP

REFERENCES:
- [Background] Morfaw F, Fundoh M, Bartoszko J, Mbuagbaw L, Thabane L. Using tocolysis in pregnant women with symptomatic placenta praevia does not significantly improve prenatal, perinatal, neonatal and maternal outcomes: a systematic review and meta-analysis. Syst Rev. 2018 Dec 27;7(1):249. doi: 10.1186/s13643-018-0923-2. PMID 30591076
- [Background] Shainker SA, Silver RM, Modest AM, Hacker MR, Hecht JL, Salahuddin S, Dillon ST, Ciampa EJ, D'Alton ME, Otu HH, Abuhamad AZ, Einerson BD, Branch DW, Wylie BJ, Libermann TA, Karumanchi SA. Placenta accreta spectrum: biomarker discovery using plasma proteomics. Am J Obstet Gynecol. 2020 Sep;223(3):433.e1-433.e14. doi: 10.1016/j.ajog.2020.03.019. Epub 2020 Mar 19. PMID 32199927
- [Background] Morlando M, Collins S. Placenta Accreta Spectrum Disorders: Challenges, Risks, and Management Strategies. Int J Womens Health. 2020 Nov 10;12:1033-1045. doi: 10.2147/IJWH.S224191. eCollection 2020. PMID 33204176
- [Background] Faraji A, Akbarzadeh-Jahromi M, Bahrami S, Gharamani S, Raeisi Shahraki H, Kasraeian M, Vafaei H, Zare M, Asadi N. Predictive value of vascular endothelial growth factor and placenta growth factor for placenta accreta spectrum. J Obstet Gynaecol. 2022 Jul;42(5):900-905. doi: 10.1080/01443615.2021.1955337. Epub 2021 Sep 24. PMID 34558384
- [Background] Seno K, Tanikawa N, Takahashi H, Ohkuchi A, Suzuki H, Matsubara S, Iwata H, Kuwayama T, Shirasuna K. Oxygen concentration modulates cellular senescence and autophagy in human trophoblast cells. Am J Reprod Immunol. 2018 Jun;79(6):e12826. doi: 10.1111/aji.12826. Epub 2018 Feb 15. PMID 29446169
- [Background] Parrish AR. Matrix Metalloproteinases in Kidney Disease: Role in Pathogenesis and Potential as a Therapeutic Target. Prog Mol Biol Transl Sci. 2017;148:31-65. doi: 10.1016/bs.pmbts.2017.03.001. Epub 2017 May 4. PMID 28662825
- [Background] Chen Y, Wang L, Bao J, Sha X, Cui L, Huang Q, Gu C, Li X, Liu H. Persistent hypoxia induced autophagy leading to invasiveness of trophoblasts in placenta accreta. J Matern Fetal Neonatal Med. 2021 Apr;34(8):1297-1303. doi: 10.1080/14767058.2019.1635582. Epub 2019 Jul 3. PMID 31269830
- [Background] Nakashima A, Tsuda S, Kusabiraki T, Aoki A, Ushijima A, Shima T, Cheng SB, Sharma S, Saito S. Current Understanding of Autophagy in Pregnancy. Int J Mol Sci. 2019 May 11;20(9):2342. doi: 10.3390/ijms20092342. PMID 31083536
- [Background] Nakashima A, Aoki A, Kusabiraki T, Cheng SB, Sharma S, Saito S. Autophagy regulation in preeclampsia: Pros and cons. J Reprod Immunol. 2017 Sep;123:17-23. doi: 10.1016/j.jri.2017.08.006. Epub 2017 Aug 26. PMID 28869810
- [Background] El-Hussieny M, Mohammed EM, Zenhom NM, Refaie MM, Okasha AM, Tawab MAE. Possible Role of TGF-beta1, MMP-2, E-CAD, beta-Catenin and Antioxidants in Pathogenesis of Placenta Accreta. Fetal Pediatr Pathol. 2021 Jun;40(3):222-232. doi: 10.1080/15513815.2020.1843574. Epub 2020 Nov 11. PMID 33172328
- [Background] Gao F, Zhou C, Qiu W, Wu H, Li J, Peng J, Qiu M, Liang C, Gao J, Luo S. Total flavonoids from Semen Cuscutae target MMP9 and promote invasion of EVT cells via Notch/AKT/MAPK signaling pathways. Sci Rep. 2018 Nov 26;8(1):17342. doi: 10.1038/s41598-018-35732-6. PMID 30478366
- [Background] Fratelli N, Prefumo F, Maggi C, Cavalli C, Sciarrone A, Garofalo A, Viora E, Vergani P, Ornaghi S, Betti M, Vaglio Tessitore I, Cavaliere AF, Buongiorno S, Vidiri A, Fabbri E, Ferrazzi E, Maggi V, Cetin I, Frusca T, Ghi T, Kaihura C, Di Pasquo E, Stampalija T, Belcaro C, Quadrifoglio M, Veneziano M, Mecacci F, Simeone S, Locatelli A, Consonni S, Chianchiano N, Labate F, Cromi A, Bertucci E, Facchinetti F, Fichera A, Granata D, D'Antonio F, Foti F, Avagliano L, Bulfamante GP, Cali G; ADoPAD (Antenatal Diagnosis of Placental Adhesion Disorders) Working Group. Third-trimester ultrasound for antenatal diagnosis of placenta accreta spectrum in women with placenta previa: results from the ADoPAD study. Ultrasound Obstet Gynecol. 2022 Sep;60(3):381-389. doi: 10.1002/uog.24889. PMID 35247287
- [Background] world health organisation. Rising rates suggest increasing numbers of medically unnecessary, potentially harmful procedures 2021 [cited 16 june 2021